CLINICAL TRIAL: NCT00873977
Title: Comparison of Three Modalities of Continuous Positive Pressure Airway Treatment for Obstructive Sleep Apnea Syndrome
Brief Title: Treatment Adherence and Outcomes in Three Modalities of Continuous Positive Airway Pressure Treatment for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Toru Oga, Medical doctor, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C-285
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Adherence; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C-flex (Active Comparator)
  Interventions: Device: CPAP (REMstar (Respironics))
- A-flex (Active Comparator)
  Interventions: Device: CPAP (REMstar (Respironics))
- Auto-CPAP (No Intervention)

INTERVENTIONS:
Device: CPAP (REMstar (Respironics)) — Pressure-relief CPAP treatment may reduce the sensation of breathing against high pressure without causing the upper airways to collapse and improve adherence.
  Other Names: REMstar (Respironics)
  Arms: A-flex; C-flex

SUMMARY:
The purpose of this study is to compare the treatment adherence and effects in three modalities of Continuous Positive Airway Pressure Treatment for Obstructive Sleep Apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder that is associated with substantial morbidity, including excessive daytime sleepiness, hypertension, and cardiovascular disease. Although Continuous Pressure Airway Pressure (CPAP) is effective treatment of objective and subjective complaints, adherence to CPAP therapy is suboptimal. Recently, pressure-relief CPAP (C-flex,A-flex; Respironics; Murrysville, PA) is available. The present study is single-blind,prospective, randomised, crossover study to compare the adherence and effects of therapy with C-flex, A-flex, and autoadjusting CPAP after 3 months of CPAP treatment.

Additionally, after 3 months of CPAP treatment, the patients who treated with C-flex and A-flex will crossovered, we will acess to change of adherence and effects of CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on admission for sleep study under the Respiratory Care and Sleep Control Medicine, Kyoto University Hospital.
* Subjects diagnosed with OSA (apnea hypopnea index >=5/hour) by overnight polysomnography.

Exclusion Criteria:

* Subjects diagnosed with CSA by overnight polysomnography.
* Subjects ever used CPAP for OSA.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
objective CPAP adherence (objective adherence are downloaded and reported by the memory card located in the CPAP device.) | 3 months

SECONDARY OUTCOMES:
subjective, objective satisfaction and complaints for CPAP therapy | 3 months
respiratory events (ie. apnea-hypopnea index) | 3 months
change of positive airway pressure | 3 months
quality of life etc. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Chin, MD,PhD, Principal Investigator — Kyoto University, Graduate School of Medicine; Yuichi Chihara, MD,PhD, Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Chihara Y, Tsuboi T, Hitomi T, Azuma M, Murase K, Toyama Y, Harada Y, Aihara K, Tanizawa K, Handa T, Yoshimura C, Oga T, Yamamoto K, Mishima M, Chin K. Flexible positive airway pressure improves treatment adherence compared with auto-adjusting PAP. Sleep. 2013 Feb 1;36(2):229-36. doi: 10.5665/sleep.2378. PMID 23372270